CLINICAL TRIAL: NCT04389801
Title: The Use of Desferal and Adjuvants for Prevention of ARDS in Hospitalised Cases Documented With Covid 19 Infection: A Randomized Controlled Trial
Brief Title: Use of Desferal for Prevention of ARDS in Hospitalised Cases Documented With Covid 19 Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hesham Al-Inany (Other)
Responsible Party: Sponsor-Investigator, Hesham Al-Inany, Prof, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0012
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19 | interventions — Deferoxamine; Injections

STUDY DESIGN:
Intervention Model Description: Desferal group An initial dose of 1000 mg should be administered at a rate NOT TO EXCEED 15 mg/kg/hr. This may be followed by 500 mg over 4 hours for two doses. Depending upon the clinical response, subsequent doses of 500 mg may be administered over 4-12 hours.
Who Masked: Participant
Masking Description: Placebo group Will receive glucose 5% over 4 hrs infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desferal (Experimental): An initial dose of 1000 mg should be administered at a rate NOT TO EXCEED 15 mg/kg/hr. This may be followed by 500 mg over 4 hours for two doses. Depending upon the clinical response, subsequent doses of 500 mg may be administered over 4-12 hours
  Interventions: Drug: Desferal 500 MG Injection
- control group (Placebo Comparator): Will receive glucose 5% over 4 hrs infusion
  Interventions: Drug: Desferal 500 MG Injection

INTERVENTIONS:
Drug: Desferal 500 MG Injection — iron chelating agent

SUMMARY:
To evaluate the efficacy of using Desferal injections for prevention of ARDS in moderate cases with fever , chest tightness and relevant chest images

DETAILED DESCRIPTION:
COVID-19 is a condition caused by a coronavirus (called SARS-CoV-2) that was first identified in late 2019. In 2020, the virus has spread to many countries around the world and neither a vaccine against the virus or specific treatment for COVID-19 has yet been developed. Recent theory showed that the severe respiratory manifestations could be due to iron toxicity which cause intense inflammation in the alveoli and hence the ground glass appearance that was seen in ragdiology imaging

Objective :

To evaluate the efficacy of using Desferal injections for prevention of ARDS in moderate cases with fever , chest tightness and relevant chest images

Randomisation:

Participants are randomly allocated to either standard care or standard care plus Desferal injection. Randomization will be done through computer generated list by principal investigator. Allocation will be determined by block randomisation, stratified by hospital. This will be carried out by an independent statistician, prior to the trial commencement, using Stata (StataCorp, College Station, TX, USA) to generate the allocation sequence. Allocations will be concealed within sequentially numbered, sealed opaque envelopes, prepared by two research assistants who are independent of the trial Blinding This study will be single blind. Doctors will not be blinded to intervention allocation due to lack of feasibility

Sample size:

Two hundred participants randomized into two groups each 100 individuals. The trial will begin as a 1:1 randomised trial Intervention Model Parallel assignment Desferal group An initial dose of 1000 mg should be administered at a rate NOT TO EXCEED 15 mg/kg/hr. This may be followed by 500 mg over 4 hours for two doses. Depending upon the clinical response, subsequent doses of 500 mg may be administered over 4-12 hours. The total amount administered should not exceed 6000 mg in 24 hours

Placebo group Will receive glucose 5% over 4 hrs infusion

Standard care :- including clexan 40, antibiotics, corticosteroids ( as anti-inflammatory agent) and hydroxychloroquine

ELIGIBILITY:
Inclusion Criteria:

* Patients positive for Covid 19 admitted to hospital with chest tightness

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Known severe hepatic impairment
* Known severe renal impairment
* Known porphyrias
* Diabetes mellitus
* Known G6PD deficiency
* Known myasthenia gravis
* Known severe psoriasis
* Known severe neurological disorders (especially those with a history of epilepsy - may lower seizure threshold)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | two weeks
  patient dies from ARDS

SECONDARY OUTCOMES:
Duration of severe symptoms | two weeks
  time to recovery

IPD SHARING:
Plan to Share IPD: Yes
email
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: five years
Access Criteria: electronic
URL: http://www.cu.edu.eg